CLINICAL TRIAL: NCT03181074
Title: Early Post-marketing Study of Daclatasvir (Daklinza) in the Treatment of Chronic Hepatitis C (CHC) in Adults
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-330
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHC patients in Mexico: patients receiving daclatasvir for the treatment of Chronic Hepatitis C at participating sentinel sites for the CNFV in Mexico
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This early post-marketing study is an observational, prospective and descriptive study of patients receiving daclatasvir for the treatment of Chronic Hepatitis C at participating sentinel sites for the CNFV in Mexico.

ELIGIBILITY:
Inclusion Criteria:

1. This study will include patients greater than or equal to 18 years of age with chronic Hepatitis C, all genotypes, including naïve and experimented (null or partial) responders, intolerant to interferon (IFN) with or without cirrhosis, HIV/HCV coinfection, and liver transplant recipients at the sentinel sites, who received at least 1 dose of daclatasvir for the treatment of chronic Hepatitis C during the specified 24-month study period.

Exclusion Criteria:

1. Subjects who received daclatasvir as part of a clinical trial.
2. Subjects who received daclatasvir for any indication other than local approved.
3. Contraindications included in the approved Mexican prescribing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic Hepatitis C who are being given daclatasvir for the treatment and cure of chronic Hepatitis C at the sentinel sites for the CNFV in Mexico. Patients will be treated according to the clinical judgment of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-10-21 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Approximately 24 months
  adverse events (AEs) on treatment with DCV in patients with chronic hepatitis C treated by doctors at participating sentinel sites for the CNFV in Mexico

SECONDARY OUTCOMES:
Distribution of Adverse Events by Age | Approximately 24 months
Distribution of Adverse Events by Gender | Approximately 24 months
Distribution of Adverse Events by Interruption or Switch of Medication | Approximately 24 months
Distribution of Adverse Events by Concomitant Medication | Approximately 24 months
Distribution of Adverse Events by Race | Approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Mexico (2):
  - Local Institution, Benito Juárez, Mexico City
  - Local Institution, Mexico City, Mexico City

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm